CLINICAL TRIAL: NCT03066440
Title: A Single-center Randomized Double Blinded Control Trial of Intravenous Fluid Content in Children With Diabetic Ketoacidosis Admitted to the Pediatric Intensive Care Unit
Brief Title: Double Blinded Randomized Control Trial of Types of IVF in Children With DKA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Shortage of potassium acetate for study intravenous fluids
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Amanda B. Hassinger, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00001394
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Ketoacidosis
Keywords: diabetic ketoacidosis; fluid management; hyperchloremia
MeSH Terms: conditions — Diabetic Ketoacidosis | interventions — Saline Solution; Sodium Chloride; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Single-center randomized double-blinded control trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The intravenous fluids administered will all have generic labeling making the study arm assignment unknown to all providers, study personnel and participants. Only the pharmacist filling the orders will known arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): Intervention: intravenous solutions containing only normal saline as the primary base during the entire treatment of diabetic ketoacidosis.
  Interventions: Drug: Normal saline
- Lactated Ringers (Experimental): Intervention: intravenous solutions containing only lactated ringers as the primary base during the entire treatment of diabetic ketoacidosis.
  Interventions: Drug: Lactated Ringers

INTERVENTIONS:
Drug: Normal saline — All intravenous fluids used in the treatment of pediatric diabetic ketoacidosis will be based in normal saline for participants in the interventional arm instead of normal saline (as given to participants in the control arm).
  Other Names: 0.9 saline
  Arms: Normal Saline
Drug: Lactated Ringers — All intravenous fluids used in the treatment of pediatric diabetic ketoacidosis will be based in lactated ringer's solution for participants in the interventional arm instead of normal saline (as given to participants in the control arm).
  Other Names: Hartmann's Solution
  Arms: Lactated Ringers

SUMMARY:
Objectives: Intravenous (IV) fluid administration is a fundamental component of diabetic ketoacidosis (DKA) treatment. Normal saline (NS), the most common IV fluid used in DKA management, contains more chloride than human blood. Excessive amounts of chloride have been shown to cause a detrimental metabolic acidosis. Other IV fluids have more physiologic chloride levels, such as lactated ringers (LR). This study will compare the rates of hyperchloremic metabolic acidosis in children treated with NS to those treated with LR to determine the effect on overall length of acidosis and length of stay in the hospital or intensive care unit.

Design: Single-center, double blinded, randomized controlled trial.

Subjects: Children aged 0 to 18 years who present with diabetic ketoacidosis and require pediatric intensive care unit admission. Patients with evidence of shock, multi-organ failure or clinically significant cerebral edema will be excluded. The projected study population will be 104 patients, 52 in each arm.

Interventions: Patients will be enrolled within 1 hour of presentation to the emergency room or pediatric intensive care unit if transferred directly from another facility. They will be randomized to receive intravenous fluids containing 0.9% saline or lactated ringers. All patients will be treated using the institutional DKA protocol with the content of the intravenous fluids being the only difference in treatment between arms. Study intervention lasts until the end of the acute management of DKA.

Planned measurements and study outcomes: The primary study outcome will be duration of metabolic acidosis. Resolution of metabolic acidosis will be defined in three ways: 1. Normalization of the ketosis; 2. Normalization of the serum pH; 3. Normalization of the serum bicarbonate level. Secondary outcomes will include length of stay in the pediatric intensive care unit and length of stay in the hospital. All outcomes will be correlated with the overall chloride load given via intravenous fluids during DKA management. Regression modelling will control for any baseline differences between the groups in regards to severity of DKA, and if newly diagnosed or poorly controlled diabetes mellitus.

DETAILED DESCRIPTION:
There have been limited prospective clinical studies in pediatrics patients examining the association of the chloride content of intravenous fluids and outcome in DKA. This prospective randomized controlled trial is being performed to compare the duration of acidosis and hospital length of stay in children with DKA who are admitted to a pediatric intensive care unit and are treated with intravenous fluids containing NS or LR. The primary study hypothesis is that use of LR will be associated with decreased duration of hyperchloremic metabolic acidosis and, therefore, shorter hospitalization than use of NS in the treatment of pediatric DKA.

Primary hypothesis: Children with diabetic ketoacidosis (DKA) who are treated with intravenous fluids containing lactated ringers (LR) will have a shorter duration of hyperchloremic metabolic acidosis after hospital admission than those treated with intravenous fluids containing normal saline (NS).

Secondary hypothesis: The duration of acidosis after hospital admission in children with DKA will be associated with length of stay in the intensive care unit and hospital.

Outcomes

Primary outcome

The primary study outcome will be duration of metabolic acidosis. Resolution of metabolic acidosis will be defined in three ways:

1. Serum ketone level <1mmol/L;
2. Venous pH > 7.3;
3. Serum bicarbonate level > 18mmol/L.

Secondary outcomes Secondary outcomes will include length of stay in the pediatric intensive care unit (PICU) and length of stay in the hospital.

Study design This is a single center, double blinded, randomized controlled trial with two treatment arms performed at a tertiary care children's hospital. Patients will be randomized within an hour of presentation to the hospital to receive DKA management using intravenous fluids containing primarily normal saline or lactated ringers. All other aspects of DKA management will be the same in each arm, per the institution protocol. Since both treatment arms involve using intravenous fluids which are considered standard of care in treating dehydration, a waiver of consent will be requested.

Recruitment methods Patients will be eligible for enrollment and randomization if they are admitted to the pediatric emergency room or pediatric intensive care unit from an outside hospital or facility with DKA and they meet inclusion criteria. Patients will be screened by emergency room personnel for eligibility and if PICU admission is determined, patients will be enrolled. If transferred directly to the pediatric intensive care unit, pediatric critical care fellow and attending physicians will be responsible for screening and enrollment 24 hours a day. Enrollment and randomization will occur within 1 hour of hospital presentation.

Enrollment will consist of assigning a randomization number at point of entry to the hospital (Emergency Room or Pediatric Intensive Care Unit) and placing the study DKA order set.

Randomization methods Upon enrollment, patients will be assigned a randomization number in sequential order from a previously generated randomization table provided by a statistician and available in the ER and PICU to study personnel. Each number will correlate with a treatment arm visible on a randomization table with coordinated treatment arm assignment available only to pharmacy personnel. Pharmacy personnel will then provide the appropriate content to the intravenous fluids with a generic label "DKA study fluids with dextrose" and "DKA study fluids without dextrose." As the fluids look identical, they would only differ visually in labelling, so standardized labelling as described here will allow all treating physicians to be blinded to treatment arm assignment.

Study Intervention All enrolled patients will be treated using the institutional DKA management protocol which is in place in the emergency room and the pediatric intensive care unit and was developed in collaboration with the endocrinology division. The only difference in the study protocol from the institutional DKA protocol is the intravenous fluid content. Please refer to study protocol schematic shown in supplement 1.

Upon admission to the ER or PICU, all eligible patients will be placed on cardiac monitors, admission DKA laboratory tests will be ordered and an initial intravenous fluid bolus of 10 ml/kg normal saline will be administered as is standard of care. These aspects of DKA management will likely be performed before study enrollment, but if not, will be identical for both arms so treatment arm assignment will not be affected. Subjects will be started on a continuous insulin infusion drip at 0.1 U/kg/hr and study intravenous fluids without dextrose at 1.5 times maintenance. Per standard of care, point of care whole blood glucose levels will be followed hourly, serum blood gases and electrolytes every 2 hours, beta-hydroxybutyrate levels every 6 hours and urine ketones every void. ER subjects will be transferred to the PICU to continue exactly the same management and laboratory schedule.

The study protocol will be used until acute management for DKA using the continuous insulin infusion is stopped. Our current practice is to convert from continuous insulin to intermittent subcutaneous insulin administration when the venous pH is equal to or greater than 7.30 and the serum bicarbonate level is equal to or greater than 15 mmol/L.

Fluid Management DKA fluid management is based on a two-bag system to maintain glucose levels between 100 and 300 mg/dL as the ketosis is corrected. The first type of intravenous fluid used has no dextrose in it to avoid worsening the initial hyperglycemia. Once the serum glucose falls below 300 mg/dL, 10% dextrose-containing fluids will be started. All intravenous fluids will contain 20millieqilivants per liter (mEq/L) of potassium acetate and 20mEq/L potassium phosphate.

Study fluid management will follow the same guidelines for rate of fluid delivery and amount of dextrose used in the standard management of patients in DKA. Bedside healthcare personnel will treat all study subjects identically regardless of treatment arm. To provide blinding to all bedside staff, intravenous fluid bags will be labelled as "DKA study fluid with dextrose" or "DKA study fluid without dextrose." All intravenous fluids used will have an electrolyte composition of 20mEq/L of potassium acetate and 20mEq/L of potassium phosphate.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 0 and 18 years
2. Diagnosis of DKA:

   1. Venous pH less than 7.25
   2. Ketonuria as confirmed on urine point-of-care testing or urinalysis
   3. Hyperglycemia (Serum glucose > 200 mg/dl)
   4. Serum bicarbonate <15 mmol/L
3. PICU admission

Exclusion Criteria:

1. Age > 18 Years
2. Physician discretion
3. Septic or hypovolemic shock
4. Signs of life-threatening cerebral edema or multi-organ failure upon presentation to the emergency room or pediatric intensive care unit
5. Enrollment time more than 1 hr since arrival to emergency room or PICU
6. Pregnancy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda B Hassinger, MD, MS, Principal Investigator — SUNY University at Buffalo
Locations (1):
- John R. Oishei Children's Hospital, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited when presenting to a tertiary care free-standing children's hospital in diabetic ketoacidosis from October 2018 to June 2021 when the study was suspended by the facility pharmacy due to a critical shortage of electrolytes for all IVF bags.
  The study was ended early in March 2024 when the pharmacy informed the study team electrolytes will not be available in a reasonable timeframe.
Pre-assignment Details: Upon enrollment, patients were randomized and treated in a double blind design
Groups:
- Normal Saline (Controls): Intravenous solutions containing only normal saline as the primary base were given during duration of treatment of diabetic ketoacidosis.
- Lactated Ringers (Intervention): Intravenous fluids containing lactated ringer's as the primary base were given during the duration of treatment of pediatric diabetic ketoacidosis.
Period: Overall Study
Arm/Group | Normal Saline (Controls) | Lactated Ringers (Intervention)
Started | 26 | 27
Completed | 25 | 24
Not Completed | 1 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Normal Saline: All intravenous fluids used in the treatment of pediatric diabetic ketoacidosis will be based in normal saline for control participants
- Lactated Ringers: All intravenous fluids used in the treatment of pediatric diabetic ketoacidosis will be based in lactated ringer's solution for participants in the interventional arm
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Lactated Ringers | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 160 [114.5 to 194] | 155.5 [130 to 187.8] | 158 [123.5 to 188.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 9 | 12 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 15 | 18 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
Admission HgbA1C [Median (Inter-Quartile Range); unit: mmol/mol] | 12.9 [10.9 to 15] | 12.8 [11.6 to 14.3] | 12.8 [11.3 to 14.4]
New onset Type 1 Diabetes [Number; unit: participants] | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Length of Acidosis
Description: Hours to pH>7.25 and normal anion gap and serum bicarbonate over 15
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Normal Saline (Controls) | Lactated Ringers (Intervention)
Number analyzed (Participants) | 25 | 24
Hours | 19.4 [11.6 to 29.1] | 19.8 [12.9 to 23.3]

2. Secondary Outcome: Length of Stay in the Pediatric Intensive Care Unit
Description: Time from admission to the emergency room or pediatric intensive care unit and transfer from the pediatric intensive care unit to the general pediatric ward
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Normal Saline (Controls) | Lactated Ringers (Intervention)
Number analyzed (Participants) | 25 | 24
days | 0.97 [0.75 to 1.40] | 1.1 [0.92 to 1.6]

3. Secondary Outcome: Length of Stay in the Hospital
Description: Time from admission to the emergency room or pediatric intensive care unit and transfer from the pediatric intensive care unit to discharge home
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Normal Saline (Controls) | Lactated Ringers (Intervention)
Number analyzed (Participants) | 25 | 24
days | 1.9 [1.2 to 2.3] | 2.0 [1.8 to 2.7]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the entirety of the participants hospital stay, up to 28 days.
Arm/Group | Normal Saline (Controls) | Lactated Ringers (Intervention)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 2/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (Controls) (N=26) | Lactated Ringers (Intervention) (N=27)
Improper Consent Obtained (Investigations) | 0 (0) | 2 (2) — Study procedure began without proper informed consent being obtained

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT03066440/Prot_SAP_000.pdf